CLINICAL TRIAL: NCT03062722
Title: Efficacy of Keyhole Approach to Carpal Tunnel Syndrome Under Ambulatory
Brief Title: Efficacy of Keyhole Approach to Carpal Tunnel Syndrome Under Ambulatory Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivan Segura Duran (Other)
Responsible Party: Sponsor-Investigator, Ivan Segura Duran, M.D., University of Guadalajara
Organization: University of Guadalajara (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI.063-2014
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Carpal Tunnel Syndrome; Entrapment Neuropathy
Keywords: microsurgical treatment; pain; dexterity; Phalen sign; functional status
MeSH Terms: conditions — Carpal Tunnel Syndrome; Charcot-Marie-Tooth Disease; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- keyhole approach (Experimental): open minimally invasive approach
  Interventions: Procedure: keyhole approach

INTERVENTIONS:
Procedure: keyhole approach — The surgical procedure was a direct microsurgical approach with a 1.5 cm incision in the thenar sulcus, under local anesthesia (3cc, 2% lidocaine) administered with an insulin needle. The keyhole approach applied to this anatomical region is based on a 1.5 cm skin incision from where the 0.5 cm dissection is completed in the subcutaneous plane in the side borders and 1cm in the distal and proximal borders. Thus, the subcutaneous phase of the dissection is completed with separation of the carpal ligament and resection of its borders. Once the transverse fibers are open, the perineural micro adhesions of the median nerve are resected and 3mm of the free borders of the carpal fibers found on the nerve are removed to avoid fibrosis. The wound is checked for hemostasis and closed in apposition with Vicryl 3-0 and a single subdermal 3-0 Nylon stitch.

SUMMARY:
Prospective controlled clinical trial in which a minimally invasive microsurgical approach was used following the keyhole principle in 55 patients and 65 hands under local anesthesia and ambulatory strategy. All patients included in the study had an average of 3 months disease course and were considered refractory to conservative treatment. Patients were evaluated with stringent inclusion criteria with the Levine severity and functional status scale with a 2 year follow-up. Descriptive outcomes on the efficiency of this procedure are reported.

DETAILED DESCRIPTION:
Prospective clinical study to analyze 55 patients with carpal tunnel syndrome treated with open minimally invasive approach in 65 hands, using local anesthesia without tourniquet and in an ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis who had neurologic exam, electromyography, cervical spine X rays showing no structural disturbances and with at least 3 months of persistent pain refractory to medical management and physical therapy.

Exclusion Criteria:

* Patients with a history of direct trauma or orthopedic lesions in the carpal region, endocrine and/or metabolic disturbances (hypothyroidism, diabetes) and those that had previous local administration of steroids were excluded.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Levine Severity Scale | 2 years follow up
  pain grades with 5 grades of intensity

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ramos Zuñiga, M.D. PhD, Principal Investigator — Universidad se Guadalajara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos-Zuniga R, Garcia-Mercado CJ, Segura-Duran I, Zepeda-Gutierrez LA. Efficacy of Keyhole Approach to Carpal Tunnel Syndrome under Ambulatory Strategy. Neurol Res Int. 2017;2017:3549291. doi: 10.1155/2017/3549291. Epub 2017 Apr 6. PMID 28484650